CLINICAL TRIAL: NCT06646965
Title: Efficacy of Family-based Dietary Counseling During Pregnancy on Gestational Weight Gain in Pregnant Women
Brief Title: Efficacy of Family-based Dietary Counseling During Pregnancy on Gestational Weight Gain in Pregnant Women in a Randomized Controlled Trial
Acronym: FAM-DIET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RC31/23/0374
Record Dates: First submitted 2024-10-15; First posted 2024-10-17 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Pregnancy; Dietetics
Keywords: Gestational weight gain; Birth weight; Recommendations; Intervention; Nutrition
MeSH Terms: conditions — Gestational Weight Gain; Birth Weight

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized, open-label clinical study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- individual dietetic follw-up (Experimental): the patient receives individual counseling (as usual clinical practice if the pregnant woman is followed by a dietetician during her pregancy).
  Interventions: Procedure: individual dietetic counseling
- family-based dietary counseling follw-up (Active Comparator): the woman and the person who shares meals with her receive family-based counseling by a dietetician during her pregancy.
  Interventions: Procedure: family-based dietetic conseling

INTERVENTIONS:
Procedure: individual dietetic counseling — only the pregnant patient receives dietetic counseling
  Arms: individual dietetic follw-up
Procedure: family-based dietetic conseling — the pregnant patient and her companion receive dietetic counseling
  Arms: family-based dietary counseling follw-up

SUMMARY:
The study aims to evaluate the efficacy of a family-based dietary monitoring during pregnancy on gestational weight gain in pregnant women. The study will be conducted as a randomized controlled trial, women will be randomly allocated into two groups: a group receiving family-based dietary monitoring, and a control group receiving individual dietary monitoring per standard recommendation.

ELIGIBILITY:
Inclusion Criteria:

Adult (+18 years old) Pregnant woman who can be accompanied by a member of the household, adult sharing at least 1 meal per day with her. Affiliated to the social security. French speaking person (read/written and spoken). Single pregnancy between 8 SA and 16 SA. Starting BMI between 18.5 and 35

Exclusion Criteria:

* Person under legal protection or guardianship
* Women suffering from a disease requiring a dietary follow-up:
* Type 1 or type 2 diabetes.
* Gestational diabetes diagnosed on the basis of fasting blood sugar.
* History of bariatric surgery.
* Eating disorders.
* Metabolic pathologies leading to special diets (phenylketonuria).
* Digestive pathologies (with an indication) with special diets
* Women who have lost more than 10% of their weight at the beginning of pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1374 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2027-06-15 (Estimated); Study Completion 2028-06-15 (Estimated)

PRIMARY OUTCOMES:
Maternal weight change | delivery
  Maternal weight change will be calculated from the difference between the weight at delivery and the pre-pregnancy weight,

SECONDARY OUTCOMES:
evaluation of BMI during pregnancy | from day 0 to delivery
  from the weight of the patient, the BMI is calculated
Weight of the baby at birth | delivery
  The weight of the child will be measured at delivery by a baby-scale measured in kilograms on the day of birth. This weight will be adjusted to the gestational age, in accordance with ARS recommendations defining weight standards according to gestational age.
The women's nutritional intake and its distribution | 16 weeks of gestation, 24 weeks of gestation, 34 of gestation, 6 months of gestation
  The women's nutritional intake and its distribution will be assessed through a food frequency questionnaire and recall from 24 hours to 16 SA (over a period of 8-16 SA). At the next two appointments during pregnancy and postpartum, a 3-day dietary survey will be conducted at 24 SA (over a period of 21- 24 SA) and 34 SA (over a period of 31-34 SA), as well as at 6 months postpartum
Screening for gestational diabetes | 16 weeks of gestation, 24 weeks of gestation, 34 weeks of gestation
  by fasting blood glucose or OGTT (orally induced glucose)
Maternal weight loss | 6 months after delivery
  Maternal weight loss will be calculated by the difference between the weight at delivery and the weight 6 months after delivery
Compliance | 24 weeks of gestation, 34 weeks of gestation, 6 months after delivery
  measured with the Goal Attainment Scaling (GAS)
Physical activity | 16 weeks of gestation, 24 weeks of gestation, 34 of gestation, 6 months of gestation
  will be measured with the Pregnancy Physical Activity Questionnaire (PPAQ)
The support of the entourage | 34 weeks of gestation, 6 months after delivery
  will be measured by the Sarason Social Support Questionnaire (SSQ6 )
Women's satisfaction with their follow-up during pregnancy | 34 weeks of gestation, 6 months after delivery
  will be assessed by means of a satisfaction survey adapted to the needs of the study at 34 days' gestation
Direct medical, non-medical and indirect costs, valued from the French Healthcare insurance | from day 0 to 6 months after delivery
  measured with the EQ-5D-5L questionnaire evaluated at 6 months after delivery (for the cost-utility analysis), the number of caesarean sections avoided (for the cost-effectiveness analysis)

CONTACTS AND LOCATIONS:
Overall Officials: Clemence ROUBLIN, Study Director — University Hospital of Toulouse
Locations (3):
- France (3):
  - Hospital of Auch, Auch
  - Clinique Rive Gauche, Toulouse
  - University Hospital of Toulouse, Toulouse